CLINICAL TRIAL: NCT05855954
Title: Application of Controlled Low Central Venous Pressure Technique in Early Intervention of Cardiac Surgery-associated Acute Kidney Injury
Brief Title: Application of CLCVP Technique in Early Intervention of CSA-AKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ClinicalTrials20230321
Record Dates: First submitted 2023-03-21; First posted 2023-05-12 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-10

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury (AKI); Controlled Low Central Venous Pressure (CLCVP); Central Venous Pressure (CVP); Postoperative Cognitive Dysfunction (POCD)
MeSH Terms: conditions — Acute Kidney Injury; Postoperative Cognitive Complications

STUDY DESIGN:
Intervention Model Description: intervention group and control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): First,20min after the end of cardiopulmonary bypass, on the basis of ensuring that the mean arterial pressure (MAP) ≥ 60mmHg, the patients will accept dorsal elevated position.
  After that, if the patient's CVP is less than 10mmHg, nitroglycerin will be pumped at 0.2ug/ (kg * min). If the patient's CVP is still greater than or equal 10mmHg, we increase the dose by 0.2ug/ (kg * min) and pump again for 5min, and the like. Until the patient's CVP is less than 10mmHg or the dose of nitroglycerin increases to 1ug/ (kg * min), the current dose is maintained until the end of surgery.
  Interventions: Combination Product: controlled low central venous pressure technique (CLCVP)
- control group (No Intervention): no intervention measures

INTERVENTIONS:
Combination Product: controlled low central venous pressure technique (CLCVP) — 20min after the end of cardiopulmonary bypass, on the basis of ensuring that the mean arterial pressure (MAP) ≥ 60mmHg, we maintain the patient's central venous pressure below 10 mmHg by adjusting the posture and pumping nitroglycerin.
  Arms: intervention group

SUMMARY:
The goal of this clinical trial is to learn about in postoperative acute kidney injury in cardiac surgery. The main questions it aims to answer are:

1. Controlled low central venous pressure (CLCVP) technique can reduce the occurrence of cardiac surgery-associated acute kidney injury (CSA-AKI) by reducing venous congestion and increasing renal perfusion pressure.
2. CLCVP technique does not increase the risk of postoperative cognitive dysfunction (POCD) during cardiac surgery.

Participants who are assigned to the intervention group will receive CLCVP technique. Specific methods are as follows: First,20min after the end of cardiopulmonary bypass, on the basis of ensuring that the mean arterial pressure (MAP) ≥ 60mmHg, the patients will accept dorsal elevated position. After that, if the patient's central venous pressure (CVP) is less than 10mmHg, nitroglycerin will be pumped at 0.2ug/ (kg * min). If the patient's CVP is still greater than or equal 10mmHg, we increase the dose by 0.2ug/ (kg * min) and pump again for 5min, and the like. Until the patient's CVP is less than 10mmHg or the dose of nitroglycerin increases to 1ug/ (kg * min), the current dose is maintained until the end of surgery.

If participants are assigned to the control group, no intervention measures will be taken.

The researchers will compare the intervention group with the control group to see the occurrence of CSA-AKI and POCD after cardiac surgery.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is a common and serious complication after cardiac surgery, which is associated with worsen prognosis including longer hospitalization, elevated mortality and morbidity and greater healthcare costs.The pathophysiological mechanisms underlying the development of AKI after cardiac surgery are complex. Venous congestion during cardiac surgery rather than hypotension is independently associated with the postoperative adverse kidney events, for both AKI within 7 days postoperative and longer-term acute kidney disease (AKD) that develops between 8- and 90-day postoperative window.Central venous pressure (CVP) is used as an indicator to quantify the degree of venous congestion, and high CVP may reflect severe venous congestion, contributing to decreased organ perfusion pressure and negatively affect renal microcirculation.

Controlled low central venous pressure (CLCVP) technique is a common and safe technique in clinical surgery.CLCVP technology has been widely used in hepatectomy, but there are few studies on its application in cardiac surgery settings. Most scholars believe that it has no adverse effects on the kidneys, while some studies suggest that it has a certain protective effect on the kidneys, but the mechanism is unclear.Actively targeting lower CVP levels using fluid restriction, reverse Trendelenburg position, vasodilators and other methods by anesthetics, can significantly reduce major intraoperative bleeding events.CLCVP technique could potentially play a role in renal protection during cardiac surgery by easing venous congestion through reduced CVP levels.

We therefore carried out a controlled randomized clinical trial to study the effect of CLCVP technique on postoperative acute kidney complications after on-pump cardiac surgery. Specifically, we tested the hypothesis that CLCVP management reduces the incidence of postoperative AKI through lower intraoperative CVP levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older, who underwent cardiac surgery (coronary artery bypass grafting (CABG), heart valve surgery, heart transplant or surgical excision of intracardiac myxoma) were eligible for analyses.

Exclusion Criteria:

* pre-existing renal insufficiency defined by presence of abnormal preoperative serum creatinine ≥ 133 μmol/L and/or preoperative diagnosis of renal insufficiency within 6 months' preoperative period.
* patients with preoperative dialysis dependence within 60 days before surgery, off-pump heart surgery, prior kidney transplantation, pregnancy, as well as those under drug therapy with nitroglycerin were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury (AKI) 1 | preoperation, Within 7 days after surgery
  Acute Kidney Injury is defined as an absolute increase in serum creatinine of ≥0. 3 mg/dL (≥26. 5 mmol/L) within 2 days or a 1. 5-fold increase in serum creatinine from baseline within 7 days, or UO <0. 5 ml/kg/h for more than 6 hours in the ICU after surgery
Acute kidney injury (AKI) 2 | one day after surgery
  Acute Kidney Injury is defined as an absolute increase in serum creatinine of ≥0. 3 mg/dL (≥26. 5 mmol/L) within 2 days or a 1. 5-fold increase in serum creatinine from baseline within 7 days, or UO <0. 5 ml/kg/h for more than 6 hours in the ICU after surgery
Acute kidney injury (AKI) 3 | three days after surgery
  Acute Kidney Injury is defined as an absolute increase in serum creatinine of ≥0. 3 mg/dL (≥26. 5 mmol/L) within 2 days or a 1. 5-fold increase in serum creatinine from baseline within 7 days, or UO <0. 5 ml/kg/h for more than 6 hours in the ICU after surgery
Acute kidney injury (AKI) 4 | 7 days after surgery
  Acute Kidney Injury is defined as an absolute increase in serum creatinine of ≥0. 3 mg/dL (≥26. 5 mmol/L) within 2 days or a 1. 5-fold increase in serum creatinine from baseline within 7 days, or UO <0. 5 ml/kg/h for more than 6 hours in the ICU after surgery

SECONDARY OUTCOMES:
Postoperative cognitive dysfunction (POCD) 1 | preoperation
  Diagnosis of postoperative POCD using MSE scales
Postoperative cognitive dysfunction (POCD) 2 | 7 days after surgery
  Diagnosis of postoperative POCD using MSE scales
Postoperative cognitive dysfunction (POCD) 3 | 30 days after surgery
  Diagnosis of postoperative POCD using MSE scales

CONTACTS AND LOCATIONS:
Overall Officials: Yali Ge, Doctor, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen L, Hong L, Ma A, Chen Y, Xiao Y, Jiang F, Huang R, Zhang C, Bu X, Ge Y, Zhou J. Intraoperative venous congestion rather than hypotension is associated with acute adverse kidney events after cardiac surgery: a retrospective cohort study. Br J Anaesth. 2022 May;128(5):785-795. doi: 10.1016/j.bja.2022.01.032. Epub 2022 Mar 4. PMID 35249707
- [Background] Lopez MG, Shotwell MS, Morse J, Liang Y, Wanderer JP, Absi TS, Balsara KR, Levack MM, Shah AS, Hernandez A, Billings FT 4th. Intraoperative venous congestion and acute kidney injury in cardiac surgery: an observational cohort study. Br J Anaesth. 2021 Mar;126(3):599-607. doi: 10.1016/j.bja.2020.12.028. Epub 2021 Feb 4. PMID 33549321
- [Background] Correa-Gallego C, Berman A, Denis SC, Langdon-Embry L, O'Connor D, Arslan-Carlon V, Kingham TP, D'Angelica MI, Allen PJ, Fong Y, DeMatteo RP, Jarnagin WR, Melendez J, Fischer M. Renal function after low central venous pressure-assisted liver resection: assessment of 2116 cases. HPB (Oxford). 2015 Mar;17(3):258-64. doi: 10.1111/hpb.12347. Epub 2014 Nov 11. PMID 25387727
- [Background] Liu TS, Shen QH, Zhou XY, Shen X, Lai L, Hou XM, Liu K. Application of controlled low central venous pressure during hepatectomy: A systematic review and meta-analysis. J Clin Anesth. 2021 Dec;75:110467. doi: 10.1016/j.jclinane.2021.110467. Epub 2021 Aug 1. PMID 34343737